CLINICAL TRIAL: NCT03515122
Title: The Swedish Spinal Cord Injury Study on Cardiopulmonary and Autonomic Impairment
Acronym: SPICA
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Collaborators: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Jan Lexell, Professor, Senior Consultant, Lund University
Other Study IDs: 2017-0765
Record Dates: First submitted 2018-03-20; First posted 2018-05-03 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Spinal Cord Injuries; Cardiovascular Diseases; Pulmonary Disease; Autonomic Dysfunction
Keywords: Epidemiology; Rehabilitation; Clinical protocols; Middle aged
MeSH Terms: conditions — Spinal Cord Injuries; Cardiovascular Diseases; Lung Diseases; Primary Dysautonomias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, plasma-EDTA, plasma-Citrate plasma li-heparin, DNA EDTA-whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Persons with Spinal cord injury (SCI): The total population of a specified group of persons with traumatic SCI will be invited to participate.
- Matched control group: A matched control group of the general population at a ratio of 3-4 to each person with SCI will be recruited from the Swedish Cardiopulmonary and Bioimage Study.

SUMMARY:
The main aim of this study is to gain an in-depth knowledge of cardiopulmonary and autonomic health consequences, and related risk factors among people with long-term high-level spinal cord injury. The result of this study will form the basis for further research to improve prevention strategies and risk prediction of cardiopulmonary disorders in people with spinal cord injury.

DETAILED DESCRIPTION:
Life expectancy for people with spinal cord injury (SCI) has increased during the 20th century as a result of improvements in health care systems and the environment. The incidence of SCI is stable and as a consequence the prevalence of SCI has increased globally leading to a growing population of persons aging with SCI. Therefore, SCI research need to focus on the physiology of aging to prevent premature cardiovascular and pulmonary diseases, which are the leading causes of death.

The disruption of sensory-, motor- and autonomic pathways causes major neurological deficits which alter the physiologic conditions. Among people with SCI above the mid-thoracic level dysfunction in pulmonary, autonomic cardiovascular regulation and emerging metabolic cardiovascular risk factors are well-known. In addition, paralysis of the abdominal and thoracic musculature causes restrictive pulmonary dysfunction, weak cough and atelectasis contributing to the mortality in SCI.

Cardiovascular disease (CVD) is more prevalent and occurs earlier in life among people with SCI compared to the general population. The increased prevalence of traditional risk factors cannot, however, fully explain these findings. Cardiovascular autonomic dysfunction has been hypothesized to contribute to the increased risk. The need for advances in risk management is therefore important as the first symptoms of coronary atherosclerosis are commonly sudden death or acute coronary syndrome. This is further complicated by the sensory loss and reduced ability to perform strenuous activities leading to asymptomatic disease as typical symptoms of exertional angina pectoris does not manifest. Risk assessment tools, such as Framingham risk score or Systematic Coronary Risk Evaluation (SCORE), are available but lack the precision in people with SCI as these tools are calibrated on the general population.

The Swedish Spinal Cord Injury Study on Cardiopulmonary and Autonomic Impairment - SPICA - was initiated to assess the effects of aging with SCI on the cardiovascular, pulmonary and autonomic systems in a cohort of middle-aged persons with long-term SCI. SPICA combines advanced imaging techniques, likely to play an important role in risk stratification of CVD and pulmonary disease in the future, with functional analyses, and generic and SCI-specific assessment tools.

The overarching aim of SPICA is to assess and extensively characterize the cardiopulmonary and autonomic health status in middle-aged persons with a severe and high-level SCI. The study will elucidate the cardiopulmonary health consequences specific to persons living with a SCI through comparison of results to matched controls. The results of SPICA will advance the investigator's knowledge in this field and thereby improve prevention strategies and risk prediction of CVD and pulmonary disorders in people with SCI.

ELIGIBILITY:
Inclusion criteria:

* Traumatic SCI
* SCI duration >5 years
* Neurological level of lesion C1-T6
* ASIA Impairment Scale A-C
* Resident in Skåne, Sweden
* No dependency of full-time ventilation support

Control group will consist of matched controls from the Swedish Cardiopulmonary and Bioimage Study's data of the general population.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The total SCI population matching the inclusion criteria in Skåne, Sweden (n=38).
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Coronary artery calcium score | Day 1
  Measures the amount of calcium in the coronary arteries from computed tomography imaging. Scores from 0 to >1000, a higher value represents a worse outcome. Value >0 indicates coronary atherosclerosis.
Intima media thickness in the carotid arteries | Day 1
  Ultrasound of carotid arteries to measure intima media thickness
Assesses atherosclerosis in the coronary arteries | Day 1
  Coronary CT Angiography
Prevalence of structural changes in the lung tissue | Day 1
  High resolution CT scan
Ectopic fat distribution | Day 1
  CT body composition of epicardium, liver, abdomen and muscle
Heart rate response to deep breathing | Day 1
  Measures electrocardiography the activity of the autonomic nervous system based on the time and frequency domain indices of heart rate variability during deep breathing.
Orthostatic blood pressure | Day 1
  Measures systolic and diastolic blood pressure changes from supine position and after 3 minutes in seating position.
Plaques in the carotid arteries | Day 1
  Ultrasound of carotid arteries to measure and characterize plaques.

SECONDARY OUTCOMES:
Questionnaire | Day 1
  self-reported health, lifestyle, social determinants, living conditions and medical history
Spinal Cord Injury Spasticity Evaluation Tool (SCI-SET) | Day 1
  Self-reported spasticity scale that measures the impact of spasticity in activities of daily living. Ranges from -105 to 105. Low values represents a worse outcome
Sense of Coherence Scale (SOC-13) | Day 1
  To assess the 3 dimensions of the SOC concept: comprehensibility (5 items), manageability (4 items), and meaningfulness (4 items). Value ranges from 13 to 91 and low values represent a worse outcome.
Hospital Anxiety and Depression Scale (HADS) | Day 1
  Screening instrument for anxiety and depression. Consists of two subscales, one for depression and one for anxiety each ranging from 0-21, high value represents a worse outcome.
Spinal Cord Independence Measure (SCIM III) | Day 1
  SCIM III comprises 19 areas of activities of daily living grouped into 3 subscales: self-care, respiratory and sphincter management, and mobility and measure self-reported activity limitation. SCIM III ranges from 0-100 and a low value represents a worse outcome.
Modified Ashworth Scale | Day 1
  Clinical examination of spasticity in specific muscles of the upper and lower extremities. The scale ranges from 0-4 with increasing scores indicating increased spasticity.
American Spinal Injury Association (ASIA) Impairment Scale | Day 1
  Measures the extent of spinal cord injury and the neurological level of injury. The extent of injury is classified as A-E. A (complete injury); B (sensory incomplete injury); C (motor incomplete injury, more than half of key muscle functions below the neurological level have a muscle grade 2 or less); D (motor incomplete injury, at least half of key muscle functions below the neurological level have a muscle grade 3 or more); E (normal sensory and motor function). i.e. from complete to normal neurological function. Thus A represents a worse outcome than E. The neurological level of injury reflects the most rostral spinal cord level with normal sensory and motor function.
Autonomic Dysfunction Following Spinal Cord Injury (ADFSCI) | Day 1
  Measures the occurrence and severity of autonomic dysreflexia (AD) and hypotension in spinal cord injury. Consists of two subscales ranging from 0-204 (AD) and 0-232 (hypotension) and a high value represents a worse outcome.
Total cholesterol | Day 1
  Analysis of venous blood sample for total cholesterol levels
High density lipoproteins (HDL) | Day 1
  Analysis of venous blood sample for total HDL-levels
Low density lipoproteins (LDL) | Day 1
  Analysis of venous blood sample for LDL-levels
Triglycerides | Day 1
  Analysis of venous blood sample for triglycerides levels
Fasting plasma glucose | Day 1
  Analysis of venous blood sample for fasting plasma glucose level
Glycated hemoglobin (HbA1c) | Day 1
  Analysis of venous blood sample for HbA1c level
high sensitive C-reactive protein (hsCRP) | Day 1
  Analysis of venous blood sample for hsCRP level
Cystatin C | Day 1
  Analysis of venous blood sample for Cystatin C level
Creatinine | Day 1
  Analysis of venous blood sample for Creatinine level
Urate | Day 1
  Analysis of venous blood sample for Urate level
Hemoglobin | Day 1
  Analysis of venous blood sample for Hemoglobin level
Erythrocytes | Day 1
  Analysis of venous blood sample for erythrocytes level
Erythrocyte volume fraction (EVF) | Day 1
  Analysis of venous blood sample for EVF level
Leukocytes | Day 1
  Analysis of venous blood sample for leukocytes level
Trombocytes | Day 1
  Analysis of venous blood sample for trombocytes level
Erythrocytes Mean Corpuscular Hemoglobin (Erc-MCH) | Day 1
  Analysis of venous blood sample for Erc-MCH level
Erythrocytes Mean Corpuscular Volume (Erc-MCV) | Day 1
  Analysis of venous blood sample for Erc-MCV level
Neutrophils | Day 1
  Analysis of venous blood sample for neutrophils level
Eosinophils | Day 1
  Analysis of venous blood sample for Eosinophils level
Basophils | Day 1
  Analysis of venous blood sample for Basophils level
Lymphocytes | Day 1
  Analysis of venous blood sample for lymphocytes level
Monocytes | Day 1
  Analysis of venous blood sample for monocytes level
Absolute glomerular filtration rate (GFR) | Day 1
  Calculated absolute GFR from Cystatin C level, body height, body weight, age and gender.
Body weight | Day 1
  Recorded in kilograms with a portable scale for wheelchairs.
Body height | Day 1
  Recorded in centimeters in supine position using a flexible measure tape
Waist circumference | Day 1
  Recorded in centimeters in supine position using a flexible measure tape
Hip circumference | Day 1
  Recorded in centimeters in supine position using a flexible measure tape
Body mass index | Day 1
  Produced by dividing the body weight in kilograms with the body height in meters to the power of two
Accelerometry | Seven days
  Measures ambulatory activity for seven days
Resting blood pressure | Day 1
  Standard resting systolic and diastolic blood pressure
Ankle-brachial index | Day 1
  Measures atherosclerosis in the lower extremities by dividing the systolic blood pressure at the ankle with the systolic blood pressure of the arm.
Ambulatory 24-hour blood pressure | Day 1
  Monitors systolic and diastolic blood pressures every 30 minutes over 24 hours
Electrocardiography | Day 1
  Standard 12-lead ECG recording
24-hour Holter-ECG | Day 1
  Monitors the heart activity
Advanced glycation endproduct (AGE) | Day 1
  Measures AGE in the skin
Spirometry | Day 1
  Dynamic spirometry
Gas diffusing capacity (DLCO) | Day 1
  Measures diffusing capacity of the lungs using the single breath method
Impulse oscillometry | Day 1
  Measures lung mechanics
Arterial stiffness | Day 1
  Estimated by pulse wave analysis
Arterial stiffness | Day 1
  Measured using pulse wave velocity

CONTACTS AND LOCATIONS:
Overall Officials: Jan Lexell, Professor, Principal Investigator — Lund University
Locations (1):
- Rehabilitation medicine Research Group, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Devivo MJ. Epidemiology of traumatic spinal cord injury: trends and future implications. Spinal Cord. 2012 May;50(5):365-72. doi: 10.1038/sc.2011.178. Epub 2012 Jan 24. PMID 22270188
- [Background] Groah SL, Charlifue S, Tate D, Jensen MP, Molton IR, Forchheimer M, Krause JS, Lammertse DP, Campbell M. Spinal cord injury and aging: challenges and recommendations for future research. Am J Phys Med Rehabil. 2012 Jan;91(1):80-93. doi: 10.1097/PHM.0b013e31821f70bc. PMID 21681060
- [Background] Warburton DE, Eng JJ, Krassioukov A, Sproule S; the SCIRE Research Team. Cardiovascular Health and Exercise Rehabilitation in Spinal Cord Injury. Top Spinal Cord Inj Rehabil. 2007 Summer;13(1):98-122. doi: 10.1310/sci1301-98. PMID 22719205
- [Background] Schilero GJ, Radulovic M, Wecht JM, Spungen AM, Bauman WA, Lesser M. A center's experience: pulmonary function in spinal cord injury. Lung. 2014 Jun;192(3):339-46. doi: 10.1007/s00408-014-9575-8. Epub 2014 Apr 11. PMID 24723067
- [Background] Bergstrom G, Berglund G, Blomberg A, Brandberg J, Engstrom G, Engvall J, Eriksson M, de Faire U, Flinck A, Hansson MG, Hedblad B, Hjelmgren O, Janson C, Jernberg T, Johnsson A, Johansson L, Lind L, Lofdahl CG, Melander O, Ostgren CJ, Persson A, Persson M, Sandstrom A, Schmidt C, Soderberg S, Sundstrom J, Toren K, Waldenstrom A, Wedel H, Vikgren J, Fagerberg B, Rosengren A. The Swedish CArdioPulmonary BioImage Study: objectives and design. J Intern Med. 2015 Dec;278(6):645-59. doi: 10.1111/joim.12384. Epub 2015 Jun 19. PMID 26096600
- [Derived] Hill M, Jorgensen S, Engstrom G, Persson M, Platonov PG, Hamrefors V, Lexell J. Cardiovascular autonomic function in middle-aged people with long-term cervical and upper thoracic spinal cord injuries. J Spinal Cord Med. 2025 May;48(3):447-460. doi: 10.1080/10790268.2024.2403791. Epub 2024 Oct 11. PMID 39392470